CLINICAL TRIAL: NCT03293498
Title: A Phase 1/2, Randomized, Observer-Blinded, Active-Controlled Trials to Evaluate the Safety and Immunogenicity of a Recombinant Trivalent Nanoparticle Influenza Vaccine With Matrix-M1 Adjuvant (NanoFlu) in Healthy Older Adults
Brief Title: Evaluation of the Safety and Immunogenicity of a Recombinant Trivalent Nanoparticle Influenza Vaccine With Matrix M-1 Adjuvant (NanoFlu)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: tNIV-E-101
Record Dates: First submitted 2017-09-19; First posted 2017-09-26 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Low dose NanoFlu - Day 0; Fluzone HD - Day 21
  Interventions: Biological: NanoFlu; Biological: Fluzone HD - Day 21
- Group B (Experimental): High dose NanoFlu - Day 0; Fluzone HD - Day 21
  Interventions: Biological: NanoFlu; Biological: Fluzone HD - Day 21
- Group C (Active Comparator): Fluzone HD - Day 0; Saline - Day 21
  Interventions: Biological: Fluzone HD - Day 0; Other: Saline - Day 21

INTERVENTIONS:
Biological: NanoFlu — Vaccine
  Arms: Group A; Group B
Biological: Fluzone HD - Day 0 — Vaccine
  Arms: Group C
Biological: Fluzone HD - Day 21 — Vaccine
  Arms: Group A; Group B
Other: Saline - Day 21 — Placebo
  Arms: Group C

SUMMARY:
This was a Phase 1/2, randomized, observer-blinded, active-controlled trial to assess the Safety and Tolerability of a Recombinant Trivalent Nanoparticle Influenza Vaccine (Tri-NIV) with Matrix M1™ Adjuvant in Healthy Older Adults ≥ 60 Years of Age

DETAILED DESCRIPTION:
Study tNIV-E-101 a randomized, observer-blinded, active-controlled trial designed to evaluate the safety and immunogenicity of Novavax's insect cell-derived, egg-free, influenza vaccine (Tri-NIV) based on recombinant HA nanoparticle antigens, representing the 3 major influenza types/subtypes recommended for inclusion in the 2017 - 2018 seasonal influenza vaccine by the World Health Organization (WHO) and the Center for Biologics Evaluation and Research (CBER) Approximately 330 eligible subjects were enrolled and randomized into 1 of 3 treatment groups Each group consisted of approximately 110 subjects total, stratified by age, gender, and history of receipt of the 2016 - 17 influenza vaccine. On Day 0, subjects in Groups A and B were administered an IM injection of NanoFlu at one of two dose levels; subjects in Group C received the preconfigured comparator (Fluzone HD) at the manufacturer's recommended dose and volume. On Day 21, all Group A and B subjects were administered a rescue injection with a licensed seasonal influenza vaccine. In contrast, all Group C subjects were administered an injection with a sterile saline placebo to maintain the trial blind. Trial follow-up for each subject spanned approximately 1 year from Day 0.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy older adults, male or female,
2. Willing and able to give informed consent prior to trial enrollment, and
3. Able to attend trial visits, comply with trial requirements, and provide reliable and complete reports of adverse events.

Exclusion Criteria:

1. Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care.

   * Asymptomatic chronic conditions or findings (eg, mild hypertension, dyslipidemia) that are not associated with evidence of end-organ damage are not exclusionary provided that they are being appropriately managed and are clinically stable (ie, unlikely to result in symptomatic illness within the time-course of this trial) in the opinion of the investigator.
   * Acute or chronic illnesses or conditions which may be reasonably predicted to become symptomatic if treatment were withdrawn or interrupted are exclusionary, even if stable.
   * Acute or chronic illnesses reasonably expected to be associated with increased risks in the event of influenza infection (eg, cardio-pulmonary diseases, diabetes mellitus, renal or hepatic dysfunction, hemoglobinopathies) are exclusionary, even if stable.
   * Note that illnesses or conditions may be exclusionary, even if otherwise stable, due to therapies used to treat them (see exclusion criteria 2, 5, 8, 9).
2. Participation in research involving investigational product (drug / biologic / device) within 45 days before planned date of first injection.
3. History of a serious reaction to prior influenza vaccination, or known allergy to constituents of influenza vaccines - including egg proteins - or polysorbate 80.
4. History of Guillain-Barré Syndrome (GBS) within 6 weeks following a previous influenza vaccine.
5. Receipt of any vaccine in the 4 weeks preceding the trial vaccination and any influenza vaccine within 6 months preceding the trial vaccination.
6. Any known or suspected immunosuppressive illness, congenital or acquired, based on medical history and/or physical examination.
7. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the trial vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
8. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the trial vaccine or during the trial.
9. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature > 38.0°C, on the planned day of vaccine administration).
10. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of trial results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
11. Known disturbance of coagulation.
12. Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax
Locations (3):
- United States (3):
  - Research Site US108, Raleigh, North Carolina
  - Research Site US106, Rocky Mount, North Carolina
  - Research Site US132, Statesville, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in a study conducted at 3 different clinical sites from September 18, 2017 to October 29, 2018.
Pre-assignment Details: Healthy older adults (≥ 60 years of age) were enrolled in the study and divided into 3 treatment groups based on gender, age, and history of 2016-17 influenza vaccine. Participants were treated with different doses of Tri-NIV Vaccine (0.3 mL,0.8mL), Fluzone HD (0.8 mL), and Placebo (0.5 mL) as Intramuscular (IM) injection into the deltoid muscle.
Groups:
- Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21: Participants received 15 µg in a 0.3 mL dose of Tri-NIV vaccine, intramuscularly, at Day 0 and received 60 µg in a 0.8 mL dose of Fluzone HD, intramuscularly, at Day 21.
- Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21: Participants received 60 µg in a 0.8 mL dose of Tri-NIV vaccine, intramuscularly, at Day 0 and received 60 µg in a 0.8 mL dose of Fluzone HD, intramuscularly, at Day 21.
- Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.: Participants received 60 µg in a 0.8 mL dose of Fluzone HD, intramuscularly, at Day 0 and received 60 µg in a 0.5 mL dose of Placebo, intramuscularly, at Day 21.
Period: Overall Study
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Started | 109 | 111 | 110
Completed | 109 | 111 | 110
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 330 participants were randomized to 1 of 3 treatment groups based on age, gender, and history of receipt of the 2016 - 17 influenza vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21. | Total
Number analyzed (Participants) | 109 | 111 | 110 | 330
Age, Customized [Count of Participants; unit: Participants]
  60 to < 75 years | 90 | 91 | 90 | 271
  ≥ 75 years | 19 | 20 | 20 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 60 | 57 | 175
  Male | 51 | 51 | 53 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 108 | 110 | 109 | 327
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 13 | 9 | 39
  White | 91 | 98 | 99 | 288
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
History of Prior Flu Vaccinations [Number; unit: participants]
  Receipt of 2016 - 17 Flu Vaccine | 95 | 94 | 93 | 282
  Receipt of Flu Vaccine in Past 3 Years | 102 | 101 | 102 | 305

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All Adverse Events (AEs), Medically Attended Adverse Events (MAAEs), Serious Adverse Events (SAEs), and Significant New Medical Conditions (SNMCs).
Description: Number of participants that reported all adverse event (AE) profile (including adverse changes in clinical laboratory parameters) ; medically-attended adverse event (MAE), serious adverse event (SAE), and significant new medical condition (SNMC) post dosing.
Time Frame: Day 0 - Day 21 post dosing
Population: Group A and B participants received different doses of the Tri-NIV vaccine on Day 0 and Fluzone HD on Day 21. Group C participants received Fluzone HD on Day 0 and Placebo on Day 21.
Measure: Number; unit: participants
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Number analyzed (Participants) | 109 | 111 | 110
participants
  MAE's | 9 | 6 | 2
  SAE's | 0 | 1 | 0
  SNMC's | 0 | 1 | 0
  All AEs (21 days post-injection) | 40 | 52 | 51

2. Primary Outcome: Number of Participants With Solicited Local and Systemic AEs
Description: Number of participants with solicited local and systemic adverse events over the 7 days post-injection
Time Frame: Day 0 - Day 6 post-dosing
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Number analyzed (Participants) | 109 | 111 | 110
participants
  Solicited Local AE's (Day 0 to Day 6) | 15 | 26 | 30
  Solicited Systemic AE's (Day 0 to Day 6) | 23 | 24 | 20

3. Primary Outcome: Geometric Mean Titers (GMT) Specific for the Hemagglutinin (HA) Receptor Binding Domains of Each of the Virus Strains Included in the NanoFlu as Measured by the Hemagglutination Inhibition (HAI) Assay.
Description: The immunogenicity of Tri-NIV at 2 different doses, and the licensed comparator Fluzone HD (Sanofi Pasteur), in healthy older adults ≥ 60 years of age, based on hemagglutination inhibition (HAI) responses to vaccine-homologous influenza A and B strains, as recommended for the 2017 - 18 Northern hemisphere vaccine, at Day 21 post-dosing expressed as GMTs.
Time Frame: Day 0 - Day 21 post dosing
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Number analyzed (Participants) | 109 | 111 | 110
titers
  Day 0 (A/Michigan/45/2015 (H1N1)) | 39 [31 to 48] | 34 [27 to 42] | 31 [25 to 38]
  Day 21 (A/Michigan/45/2015 (H1N1)) | 95 [75 to 121] | 130 [102 to 166] | 139.1 [112 to 174]
  Day 0 (A/HongKong/4801/2014 (H3N2) ) | 26 [21 to 33] | 21 [17 to 27] | 26 [21 to 33]
  Day 21 (A/HongKong/4801/2014 (H3N2) ) | 62 [48 to 79] | 75 [59 to 94] | 94 [74 to 119]
  Day 0 (B/Brisbane/60/2008 (Victoria Lineage)) | 19 [15 to 23] | 18 [15 to 22] | 15 [12 to 17]
  Day 21 (B/Brisbane/60/2008 (Victoria Lineage)) | 24 [20 to 30] | 29 [24 to 35] | 37 [31 to 46]
  Day 0 (A/California/07/2009 (H1N1)) | 65 [53 to 80] | 59 [48 to 73] | 52 [42 to 64]
  Day 21 (A/California/07/2009 (H1N1) ) | 143 [116 to 176] | 194 [156 to 242] | 206 [169 to 222]
  Day 0 (A/Texas/50/2012 (H3N2) ) | 197 [155 to 251] | 160 [123 to 207] | 196 [151 to 253]
  Day 21 (A/Texas/50/2012 (H3N2) ) | 429 [352 to 523] | 485 [397 to 592] | 470 [382 to 577]
  Day 0 (A/Switzerland/9715293/2013 (H3N2)) | 65 [50 to 83] | 55 [43 to 71] | 60 [47 to 78]
  Day 21 (A/Switzerland/9715293/2013 (H3N2)) | 159 [128 to 198] | 187 [150 to 234] | 151 [122 to 188]

4. Primary Outcome: Geometric Mean Ratio (GMR) Specific for the HA Receptor Binding Domains of Each of the Virus Strains Included in the NanoFlu as Measured by the HAI Assay.
Description: The immunogenicity of Tri-NIV at 2 different doses, and the licensed comparator Fluzone HD (Sanofi Pasteur), in healthy older adults ≥ 60 years of age, based on hemagglutination inhibition (HAI) responses to vaccine-homologous influenza A and B strains, as recommended for the 2017 - 18 Northern hemisphere vaccine, at Day 21 post-dosing expressed as GMR.
Time Frame: Day 0 - Day 21 post dosing
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Number analyzed (Participants) | 109 | 111 | 110
Ratio
  Day 21 (A/Michigan/45/2015 (H1N1)) | 2.47 [2.05 to 2.98] | 3.86 [3.07 to 4.85] | 4.55 [3.60 to 5.75]
  Day 21 (A/HongKong/4801/2014 (H3N2) ) | 2.35 [1.94 to 2.84] | 3.49 [2.78 to 4.37] | 3.57 [2.87 to 4.45]
  Day 21 (B/Brisbane/60/2008 (Victoria Lineage)) | 1.30 [1.16 to 1.44] | 1.57 [1.39 to 1.78] | 2.56 [2.10 to 3.11]
  Day 21 (A/California/07/2009 (H1N1) ) | 2.20 [1.87 to 2.59] | 3.29 [2.67 to 4.05] | 3.94 [3.16 to 4.92]
  Day 21 (A/Texas/50/2012 (H3N2) ) | 2.17 [1.83 to 2.58] | 3.04 [2.48 to 3.72] | 2.40 [2.01 to 2.87]
  Day 21 (A/Switzerland/9715293/2013 (H3N2)) | 2.46 [2.04 to 2.95] | 3.38 [2.72 to 4.21] | 2.51 [2.08 to 3.02]

5. Primary Outcome: Seroconversion Rate (SCR) Specific for the HA Receptor Binding Domains of Each of the Virus Strains Included in the NanoFlu as Measured by the HAI Assay.
Description: The immunogenicity of Tri-NIV at 2 different doses, and the licensed comparator Fluzone HD (Sanofi Pasteur), in healthy older adults ≥ 60 years of age, based on hemagglutination inhibition (HAI) responses to vaccine-homologous influenza A and B strains, as recommended for the 2017 - 18 Northern hemisphere vaccine, at Day 21 post-dosing expressed as SCRs.
Time Frame: Day 0 - Day 21 post dosing
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Number analyzed (Participants) | 109 | 111 | 110
participants
  Day 21 (A/Michigan/45/2015 (H1N1)) | 34 | 49 | 54
  Day 21 (A/HongKong/4801/2014 (H3N2) ) | 24 | 34 | 43
  Day 21 (B/Brisbane/60/2008 (Victoria Lineage)) | 5 | 13 | 29
  Day 21 (A/California/07/2009 (H1N1) ) | 24 | 45 | 53
  Day 21 (A/Texas/50/2012 (H3N2) ) | 21 | 38 | 29
  Day 21 (A/Switzerland/9715293/2013 (H3N2)) | 28 | 43 | 30

6. Primary Outcome: Number of Participants With Seroprotection Specific for the HA Receptor Binding Domains of Each of the Virus Strains Included in the NanoFlu as Measured by the HAI Assay.
Description: The immunogenicity of Tri-NIV at 2 different doses, and the licensed comparator Fluzone HD (Sanofi Pasteur), in healthy older adults ≥ 60 years of age, based on hemagglutination inhibition (HAI) responses to vaccine-homologous influenza A and B strains, as recommended for the 2017 - 18 Northern hemisphere vaccine, at Day 21 post-dosing expressed as SPRs.
  Seroprotection rate (SPR) - defined as the number of subjects with an HAI titer ≥ 1:40.
Time Frame: Day 0 - Day 21 post dosing
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Number analyzed (Participants) | 109 | 111 | 110
participants
  Day 0 (A/Michigan/45/2015 (H1N1)) | 65 | 63 | 57
  Day 21 (A/Michigan/45/2015 (H1N1)) | 93 | 96 | 98
  Day 0 (A/HongKong/4801/2014 (H3N2) ) | 51 | 45 | 45
  Day 21 (A/HongKong/4801/2014 (H3N2) ) | 76 | 79 | 89
  Day 0 (B/Brisbane/60/2008 (Victoria Lineage)) | 31 | 30 | 19
  Day 21 (B/Brisbane/60/2008 (Victoria Lineage)) | 42 | 53 | 57
  Day 0 (A/California/07/2009 (H1N1) ) | 80 | 77 | 74
  Day 21 (A/California/07/2009 (H1N1) ) | 98 | 102 | 104
  Day 0 (A/Texas/50/2012 (H3N2) ) | 98 | 96 | 98
  Day 21 (A/Texas/50/2012 (H3N2) ) | 109 | 110 | 108
  Day 0 (A/Switzerland/9715293/2013 (H3N2)) | 79 | 71 | 73
  Day 21 (A/Switzerland/9715293/2013 (H3N2)) | 101 | 103 | 100

7. Secondary Outcome: Geometric Mean Titers (GMT) Specific for the HA Receptor Binding Domains of at Least 2 Historic A Virus Strains (One H1N1 and One H3N2) as Measured by the HAI Assay
Description: The immunogenicity of Tri-NIV at 2 different doses and the licensed comparator Fluzone HD (Sanofi Pasteur) based on hemagglutination inhibition (HAI) responses to at least 2 historic and/or drifted A virus strains (one H1N1 and one H3N2) expressed as GMTs.
Time Frame: Day 0 - Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Number analyzed (Participants) | 109 | 111 | 110
titers
  A/Michigan/45/2015 (H1N1) : Day 0 | 69 [61 to 78] | 66 [59 to 74] | 65 [58 to 74]
  A/Michigan/45/2015 (H1N1): Day 21 | 146 [120 to 178] | 210 [171 to 258] | 171 [141 to 206]
  A/HongKong/4801/2014 (H3N2) : Day 0 | 60 [53 to 69] | 58 [51 to 66] | 62 [53 to 74]
  A/HongKong/4801/2014 (H3N2) : Day 21 | 127 [103 to 157] | 159 [126 to 201] | 116 [91 to 147]

8. Secondary Outcome: Geometric Mean Ratio (GMR) Specific for the HA Receptor Binding Domains of at Least 2 Historic A Virus Strains (One H1N1 and One H3N2) as Measured by the HAI Assay
Description: The immunogenicity of Tri-NIV at 2 different doses and the licensed comparator Fluzone HD (Sanofi Pasteur) based on hemagglutination inhibition (HAI) responses to at least 2 historic and/or drifted A virus strains (one H1N1 and one H3N2) expressed as GMRs.
Time Frame: Day 0 - Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Number analyzed (Participants) | 109 | 111 | 110
Ratio
  A/Michigan/45/2015 (H1N1) : Day 21 | 2.13 [1.83 to 2.48] | 3.17 [2.61 to 3.85] | 2.61 [2.21 to 3.09]
  A/HongKong/4801/2014 (H3N2) : Day 21 | 2.10 [1.75 to 2.53] | 2.74 [2.22 to 3.38] | 1.85 [1.56 to 2.20]

9. Secondary Outcome: Seroconversion Rate (SCR) Specific for the HA Receptor Binding Domains of at Least 2 Historic A Virus Strains (One H1N1 and One H3N2) as Measured by the HAI Assay
Description: The immunogenicity of Tri-NIV at 2 different doses and the licensed comparator Fluzone HD (Sanofi Pasteur) based on hemagglutination inhibition (HAI) responses to at least 2 historic and/or drifted A virus strains (one H1N1 and one H3N2) expressed as SCRs.
Time Frame: Day 0 - Day 21
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Number analyzed (Participants) | 109 | 111 | 110
participants
  A/Michigan/45/2015 (H1N1): Day 21 | 27 [17.0 to 34.0] | 45 [31.6 to 50.7] | 40 [27.7 to 46.5]
  A/Michigan/45/2015 (H1N1) : Day 21 | 29 [18.6 to 35.9] | 38 [25.7 to 44.2] | 25 [15.4 to 32.0]

10. Secondary Outcome: Number of Participants With Seroprotection Specific for the HA Receptor Binding Domains of at Least 2 Historic A Virus Strains (One H1N1 and One H3N2) as Measured by the HAI Assay
Description: The immunogenicity of Tri-NIV at 2 different doses and the licensed comparator Fluzone HD (Sanofi Pasteur) based on hemagglutination inhibition (HAI) responses to at least 2 historic and/or drifted A virus strains (one H1N1 and one H3N2) expressed as SPRs.
  Seroprotection rate (SPR) - defined as the percentage of subjects with an HAI titer ≥ 1:40.
Time Frame: Day 0 - Day 21
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Number analyzed (Participants) | 109 | 111 | 110
percentage of participants
  A/Michigan/45/2015 (H1N1) : Day 0 | 99.1 [95.0 to 100.0] | 98.2 [93.6 to 99.8] | 97.2 [92.2 to 99.4]
  A/Michigan/45/2015 (H1N1) : Day 21 | 100.0 [96.7 to 100.0] | 100 [96.7 to 100.0] | 99.1 [95.0 to 100.0]
  A/HongKong/4801/2014 (H3N2) : Day 0 | 97.2 [92.2 to 99.4] | 96.4 [91.0 to 99.0] | 90.8 [83.8 to 95.5]
  A/HongKong/4801/2014 (H3N2) : Day 21 | 100.0 [96.7 to 100.0] | 98.2 [93.6 to 99.8] | 94.5 [88.4 to 98.0]

11. Secondary Outcome: Geometric Mean Titers (GMT) for Neutralizing Antibody Titers Specific for the Virus Strains Included in NanoFlu and the Fluzone HD Comparator, as Well as Selected Historical A Strains, as Measured by a Microneutralization Assay.
Description: The immunogenicity of Tri-NIV at 2 different doses, and the licensed comparator Fluzone HD (Sanofi Pasteur), based on microneutralization (MN) responses to vaccine-homologous and historic and/or drifted influenza A strains, and the vaccine-homologous B/Victoria lineage strain, at Day 21 post-dosing expressed as GMTs.
Time Frame: Day 0 - Day 21 post dosing
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Number analyzed (Participants) | 109 | 111 | 110
titers
  Day 0 (A/Switzerland/9715293/2013 (H3N2)) | 1696 [1292 to 2227] | 1258 [954 to 1658] | 1400 [1046 to 1873]
  Day 21 (A/Switzerland/9715293/2013 (H3N2)) | 4419 [3391 to 5758] | 5223 [3997 to 6824] | 3011 [2268 to 3997]
  Day 0 (A/Texas/50/2012 (H3N2)) | 3660 [2803 to 4778] | 2768 [2142 to 3577] | 3307 [2484 to 4402]
  Day 21 (A/Texas/50/2012 (H3N2)) | 9204 [7165 to 11822] | 10495 [8213 to 13410] | 8383 [6409 to 10964]
  Day 0 (A/Singapore/INFIMH-16-0019/2016 (H3N2) | 587 [461 to 748] | 437 [349 to 547] | 489 [367 to 651]
  Day 21 (A/Singapore/INFIMH-16-0019/2016 (H3N2) | 1469 [1113 to 1940] | 1640 [1254 to 2146] | 1905 [1434 to 2531]
  Day 0 (A/Michigan/45/2015 (H1N1)) | 411 [327 to 516] | 342 [269 to 436] | 334 [259 to 432]
  Day 21 (A/Michigan/45/2015 (H1N1)) | 1414 [1070 to 1868] | 2005 [1485 to 2708] | 1741 [1313 to 2309]
  Day 0 (A/HongKong/4801/2014 (H3N2) ) | 1239 [957 to 1605] | 891 [698 to 1137] | 1081 [816 to 1433]
  Day 21 (A/HongKong/4801/2014 (H3N2) ) | 3359 [2577 to 4378] | 3791 [2906 to 4944] | 4455 [3426 to 5793]
  Day 0 (B/Brisbane/60/2008 (Victoria Lineage)) | 167 [129 to 216] | 174 [137 to 220] | 154 [124 to 193]
  Day 21 (B/Brisbane/60/2008 (Victoria Lineage)) | 287 [228 to 361] | 354 [285 to 439] | 425 [341 to 529]

12. Secondary Outcome: Geometric Mean Ratio (GMR) for Neutralizing Antibody Titers Specific for the Virus Strains Included in NanoFlu and the Fluzone HD Comparator, as Well as Selected Historical A Strains, as Measured by a Microneutralization Assay.
Description: The immunogenicity of Tri-NIV at 2 different doses, and the licensed comparator Fluzone HD (Sanofi Pasteur), based on microneutralization (MN) responses to vaccine-homologous and historic and/or drifted influenza A strains, and the vaccine-homologous B/Victoria lineage strain, at Day 21 post-dosing expressed as GMRs.
Time Frame: Day 0 - Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Number analyzed (Participants) | 109 | 111 | 110
Ratio
  Day 21 (A/Switzerland/9715293/2013 (H3N2)) | 2.61 [2.13 to 3.19] | 4.15 [3.25 to 5.31] | 2.15 [1.82 to 2.55]
  Day 21 (A/Texas/50/2012 (H3N2)) | 2.51 [2.04 to 3.10] | 3.79 [3.05 to 4.72] | 2.53 [2.09 to 3.07]
  Day 21 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 2.50 [1.99 to 3.15] | 3.76 [2.98 to 4.74] | 3.90 [3.09 to 4.92]
  Day 21: A/Michigan/45/2015 (H1N1) | 3.44 [2.74 to 4.33] | 5.86 [4.45 to 7.72] | 5.21 [3.94 to 6.89]
  Day 21: A/HongKong/4801/2014 (H3N2) | 2.71 [2.20 to 3.33] | 4.25 [3.34 to 5.42] | 4.12 [3.26 to 5.20]
  Day 21: B/Brisbane/60/2008 (Victoria Lineage) | 1.72 [1.48 to 2.00] | 2.03 [1.70 to 2.43] | 2.75 [2.19 to 3.47]

13. Secondary Outcome: Seroconversion Rate (SCR) for Neutralizing Antibody Titers Specific for the Virus Strains Included in NanoFlu and the Fluzone HD Comparator, as Well as Selected Historical A Strains, as Measured by a Microneutralization Assay.
Description: The immunogenicity of Tri-NIV at 2 different doses, and the licensed comparator Fluzone HD (Sanofi Pasteur), based on microneutralization (MN) responses to vaccine-homologous and historic and/or drifted influenza A strains, and the vaccine-homologous B/Victoria lineage strain, at Day 21 post-dosing expressed as SPRs.
Time Frame: Day 0 - Day 21
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
Number analyzed (Participants) | 109 | 111 | 110
participants
  Day 21 (A/Switzerland/9715293/2013 (H3N2)) | 22 [13.1 to 29.0] | 45 [31.6 to 50.7] | 20 [11.6 to 26.9]
  Day 21 (A/Texas/50/2012 (H3N2)) | 26 [16.2 to 33.0] | 47 [33.3 to 52.5] | 28 [17.8 to 34.9]
  Day 21 (A/Singapore/INFIMH-16-0019/2016 (H3N2) | 27 [17.0 to 34.0] | 38 [25.7 to 44.2] | 43 [30.2 to 49.3]
  Day 21: A/Michigan/45/2015 (H1N1) | 33 [21.8 to 39.8] | 53 [38.6 to 57.9] | 50 [36.3 to 55.7]
  Day 21: A/HongKong/4801/2014 (H3N2) | 28 [17.8 to 34.9] | 43 [29.9 to 48.9] | 48 [34.5 to 53.9]
  Day 21: B/Brisbane/60/2008 (Victoria Lineage) | 13 [6.5 to 19.5] | 18 [10.0 to 24.6] | 23 [13.9 to 30.0]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Serious Adverse Events Other (Not Including Serious) Adverse Events
Arm/Group | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21.
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/111 | 0/110
Serious Adverse Events (participants affected / at risk) | 7/109 | 11/111 | 8/110
Other Adverse Events (participants affected / at risk) | 32/109 | 27/111 | 28/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 (N=109) | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 (N=111) | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21. (N=110)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2)
COLITIS MICROSCOPIC (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1)
BETA HAEMOLYTIC STREPTOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PELVIC ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SEROMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
CERVICAL RADICULOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A- Participants Received Low Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 (N=109) | Group B- Participants Received High Dose Tri-NIV Vaccine at Day 0 and Received Fluzone HD at Day 21 (N=111) | Group C - Participants Received Fluzone HD at Day 0 and Received Dose of Placebo at Day 21. (N=110)
BRONCHITIS (Infections and infestations) | 11 (11) | 9 (10) | 6 (6)
SINUSITIS (Infections and infestations) | 4 (4) | 5 (5) | 7 (7)
BLOOD PRESSURE SYSTOLIC INCREASED (Investigations) | 11 (11) | 4 (4) | 8 (8)
HEADACHE (Nervous system disorders) | 2 (3) | 7 (8) | 1 (1)
HYPERTENSION (Vascular disorders) | 4 (4) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT03293498/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT03293498/SAP_001.pdf